CLINICAL TRIAL: NCT00680134
Title: An Open Label, Multi-center Study To Evaluate The Safety And Efficacy Of Topically Applied An2690 1% And 5% Solutions For The Treatment Of Adult Subjects With Onychomycosis Of The Great Toenail
Brief Title: Safety and Efficacy Evaluation of Topically Applied AN2690 Solutions for Subjects With Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: AN2690-ONYC-203; C3371007 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group/Cohort 1 (Experimental): AN2690 1% Solution (30 subjects)
  Interventions: Drug: AN2690
- Group/Cohort 2 (Experimental): AN2690 5% Solution (30 subjects)
  Interventions: Drug: AN2690

INTERVENTIONS:
Drug: AN2690 — AN2690 1% Solution, once daily for 180 days
  Arms: Group/Cohort 1
Drug: AN2690 — AN2690 5% Solution, once daily for 30 days; 3x weekly for 150 days
  Arms: Group/Cohort 2

SUMMARY:
The purpose of the study is to determine the safety and efficacy of 1% and 5% AN2690 solutions in the treatment of distal, subungual onychomycosis of the great toenail.

DETAILED DESCRIPTION:
The first group of 30 protocol-qualified subjects will be assigned to Treatment Group 1 and given 1% AN2690 Solution. The second group of 30 protocol-qualified subjects will be assigned to Treatment Group 2 and given 5% AN2690 Solution.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed, signed informed consent approved by Institutional Review Board/Ethics Committee
* A signed Health Insurance Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of subject's individually identifiable health information for those enrolled in the United States of America
* Male or female subjects of any race 18 -65 years of age
* Subjects with a diagnosis of onychomycosis of at least one great toenail and with a positive KOH wet mount and a positive fungal culture for dermatophyte species
* Onychomycosis involving 20-60% of the affected great toenail as determined at baseline (Day1) by visual inspection after the nail has been trimmed
* The combined thickness of the distal nail plate and the associated hyperkeratotic nail bed <3 mm
* Affected great toenail to be treated is capable of re-growth as documented by history or recent observation of at least 2 mm of growth

Exclusion Criteria:

* Females of childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study
* Subjects unwilling to refrain from the use of nail cosmetics such as clear and or colored nail lacquers from the screening visit until the end of the study
* Subjects with chronic moccasin type of T. pedis
* Subjects with a history of having failed any previous topical antifungal therapy for their onychomycosis
* Diabetes mellitus requiring treatment other than diet and exercise
* Subjects that have not undergone the specified washout period(s) for the following topical preparations or subjects who require the concurrent use of any of the following topical medications:

  1. Topical antifungal applied to toenails (does not include antifungals for treatment of T. pedis): 12 weeks
  2. Anti-inflammatories, corticosteroids, topical immunomodulators (in the treatment area): 2 weeks
* Subjects that have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

  1. Corticosteroids (including intramuscular injections): 2 weeks
  2. Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophyte species: 24 weeks
  3. Systemic immunomodulators: 4 weeks
* Treatment of any type for cancer within the last 6 months
* History of any significant internal disease
* Subjects with a medical history of current or past psoriasis of the skin and/or nails
* Concurrent lichen planus
* Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure
* Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated
* AIDS or AIDS related complex
* History of street drug or alcohol abuse
* Any subject not able to meet the study attendance requirements
* Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06-30 (Actual); Primary Completion 2007-08-31 (Actual); Study Completion 2007-08-31 (Actual)

PRIMARY OUTCOMES:
Complete or partial clinical evidence of great toenail clearance or at least 2 mm of fungal clear linear great toenail growth plus a negative fungal culture from the treatment targeted toenail at the End-of-treatment (Day 180) | Day 180

SECONDARY OUTCOMES:
Evaluations of mycological response, changes from baseline linear toenail growth, proportion of subjects who are successful "Complete Responders" | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Bryan, Texas
  - Endeavor Clinical Trials, PA & San Antonio Podiatry Associates, PC, San Antonio, Texas